CLINICAL TRIAL: NCT05374837
Title: The Impact and Implementation of a Mobile Messaging Intervention to Improve Infant and Young Child Nutrition in Senegal
Brief Title: Mobile Messaging for Improved Nutrition
Acronym: IIMAANJE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Shauna Downs, PhD MS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2021000819; 1R21HD105067-01 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-16 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Diet, Healthy; Anemia
Keywords: Senegal; Infant and young child feeding
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Cluster-randomized control trial. Please note that enrollment number reflects the number of triads included in the study.
Masking Description: Given the nature of the intervention, it will not be possible to mask the treatment group at endline data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will not receive any intervention. After the endline data collection is completed, the intervention will be delivered to the control group.
- Infant and young child feeding (IYCF) voice messaging intervention (Experimental): The voice messaging intervention group will receive voice/text messages for a period of 16 weeks.
  Interventions: Behavioral: Infant and young child feeding voice messaging intervention

INTERVENTIONS:
Behavioral: Infant and young child feeding voice messaging intervention — A mobile voice and text messaging intervention aimed at improving IYCF practices will be delivered to mothers and fathers with young children (6-23 months). A total of 16 voice and text message, with the same content, will be sent over a 16-week period (1 voice + 1 text messages (with same content) per week x 16 weeks). Two types of messages will be included: 1) eight scripted and 2) eight unscripted messages from positive deviants. The content of the messages include: breastfeeding until two years of age, consuming a variety of foods within a given meal, the consistency of porridge (thick rather than thin), limiting sweets and fried foods, the importance of animal source foods, consuming vitamin A rich fruits and vegetables, consuming leafy greens, handwashing and feeding infants and young children fruits and vegetables produced by the household.
  Arms: Infant and young child feeding (IYCF) voice messaging intervention

SUMMARY:
This project will examine the impact of an infant and young child feeding (IYCF) voice messaging intervention delivered to mothers and fathers in Senegal on the consumption of a minimum acceptable diet and anemia prevalence in their children.

DETAILED DESCRIPTION:
This is a cluster-randomized control trial (cRCT) conducted with 488 mother, father, and child triads in 104 villages in three regions in Senegal: Thies, Diourbel and Fatick. Mothers and fathers in the experimental group will receive 16 voice and text messages over the course of 16 weeks. One voice and 1 text message with the same content will be sent per week over the 16 week period. We will include eight scripted messages which have previously been piloted. We will also include eight unscripted messages from positive deviants from communities similar to our study population that were included in our pilot study. A text message with the same content as the voice message will be sent to each triad mother and father to increase the reach of the intervention. We will conduct baseline and endline assessments of infant and young child feeding practices in both the experimental and control groups. Primary outcomes will include the prevalence of anemia and minimum acceptable diet in children. Minimum acceptable diet is an indicator of dietary diversity and a proxy for nutrient adequacy. Secondary outcomes include the frequency of consuming key foods targeted in the intervention over the previous 7 days and infant and young child feeding indicators of complementary feeding of the child. In addition, infant and young child feeding knowledge, beliefs, and norms (of mothers and fathers in triads) and intentions (of mothers in triads) will be included as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Thies, Diourbel or Fatick regions of Senegal
* Household is member of village farming group
* Mothers and fathers (or caregivers) that have a child 6-19 months at baseline
* Mothers and fathers (or caregivers) that are 18 years or older
* Mothers and fathers (or caregivers) have the ability and mental capacity to consent to their participation
* Mother/father (or male/female caregivers) have access to mobile phone
* Child between 6-19 months at baseline

Exclusion Criteria:

-Does not meet study inclusion criteria

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shauna Downs, Principal Investigator — Rutgers School of Public Health
Locations (1):
- Institut de Recherche en Santé de Surveillance Epidemiologique et de Formation, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No
Access to the study database will be available for educational, research and non-profit purposes. All data to be shared will be stripped of any potentially identifying information. Data will be made available through written request to the PIs. A brief analysis plan and data request will be required and reviewed by the PI for approval of data sharing. When requests are approved data will be sent electronically in password protected files. The final dataset will be available in a cvs file.

REFERENCES:
- [Derived] Downs SM, Gueye D, Sall M, Ndoye B, Sarr NN, Sarr M, Mboup S, Alam NA, Diouf A, Merchant EV, Sackey J. The impact and implementation of an mHealth intervention to improve infant and young child feeding in Senegal: IIMAANJE protocol for a cluster randomized control trial. Front Public Health. 2023 Sep 25;11:1258963. doi: 10.3389/fpubh.2023.1258963. eCollection 2023. PMID 37818304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited triads (mother, father and child) for this study. The intervention was delivered to mothers and fathers in the triad and the study outcomes were primarily measured in the child.
Pre-assignment Details: The enrollment number reflects the number of triads (child, mother/primary female caregiver, and father/primary male caregiver) that were enrolled in the study. The numbers started and completed reflect the individual child, mother, and father participants.
Units Other Than Participants: Village
Period: Overall Study
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Started | 455; 52 Village (205 mothers; 205 children; and 45 fathers were included at baseline.) | 632; 52 Village (283 mothers; 283 children; and 66 fathers were included at baseline)
Child Participants Started Study | 205; 52 Village | 283; 52 Village
Mother Participants Started Study | 205; 52 Village | 283; 52 Village
Father Participants Started Study | 45; 52 Village | 66; 52 Village
Child Participants Completed the Study | 205; 52 Village | 283; 52 Village
Mother Participants Completed the Study | 205; 52 Village | 283; 52 Village
Father Participants Completed the Study | 28; 52 Village | 48; 52 Village
Completed | 438; 52 Village (205 mothers; 205 children; and 28 fathers completed endline) | 614; 52 Village (283 mothers; 283 children; and 48 fathers completed endline)
Not Completed | 17; 0 Village | 18; 0 Village
Not completed — Lost to Follow-up | 17 | 18

BASELINE CHARACTERISTICS:
Population: The study population is triads (mother, father, child). Some baseline population characteristics were collected for the triad (race/ethnicity, region) and others are specific to the mother, father, or child. 205 mothers; 205 children; and 45 fathers were included at baseline.
Units Other Than Participants: Villages
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention | Total
Number analyzed (Participants) | 455 | 632 | 1087
Number analyzed (Villages) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: Months of child] — The age of child is in months. Population: These numbers reflect solely the number of children in the triads.
  Months of child
    number analyzed (Participants) | 205 | 283 | 488
    Child | 12.3 (4.6) | 11.6 (4.1) | 11.9 (4.3)
Age, Continuous [Mean (Standard Deviation); unit: Years of mother] — Age of mother included in triad Population: These numbers solely include the mothers in the triads.
  Years of mother
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 28.67 (8.06) | 27.76 (7.45) | 28.15 (7.72)
Age, Continuous [Mean (Standard Deviation); unit: Years of father] — Age of father included in triad Population: Few of the fathers included in the triad were available (because they were working in farming fields or working outside the household in other occupations) to complete the surveys asking about their infant and young child feeding knowledge, attitudes and beliefs. However, these fathers still received the intervention (if in the experimental group).
  Years of father
    number analyzed (Participants) | 45 | 66 | 111
    (all) | 42.67 (8.18) | 41.89 (9.55) | 42.21 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of child included in triad Population: The different rows present the sex of children participants, mother participants, and father participants.
  Participants
    Child participants: number analyzed (Participants) | 205 | 283 | 488
    Child participants: Female | 92 | 145 | 237
    Child participants: Male | 113 | 138 | 251
    Mother participants: number analyzed (Participants) | 205 | 283 | 488
    Mother participants: Female | 205 | 283 | 488
    Mother participants: Male | 0 | 0 | 0
    Father participants: number analyzed (Participants) | 45 | 66 | 111
    Father participants: Female | 0 | 0 | 0
    Father participants: Male | 45 | 66 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity of triad. Data were collected at the triad household level. We did not collect data separately for mothers, fathers, and child. Population: Ethnicity was measured at the triad/household level. We only report ethnicity for the triad and not for children, mother, and father participants separately.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Ethnicity of triad/household: Wolof/Lebou | 147 | 194 | 341
    Ethnicity of triad/household: Pular/Toucouleur | 13 | 6 | 19
    Ethnicity of triad/household: Serere | 39 | 75 | 114
    Ethnicity of triad/household: Diola | 2 | 0 | 2
    Ethnicity of triad/household: Manding/Soce | 2 | 4 | 6
    Ethnicity of triad/household: Other ethnicity | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants] — Region of the triad. Data were collected at the triad household level. We did not collect data separately for mothers, fathers, and child. All participants are from Senegal. Population: Data were captured at the triad level.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Senegal | 205 | 283 | 488
Child's mother's highest education level completed [Count of Participants; unit: Participants] — This is a measure of the child's mother's highest level of education completed. Population: This measure was only for mothers included in the study (n=205 in control; n=283 in experimental group)
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Primary school | 42 | 66 | 108
    Secondary school | 33 | 45 | 78
    University | 5 | 4 | 9
    Did not attend formal school | 125 | 168 | 293
Prevalence of child anemia [Count of Participants; unit: Participants] — Hemocue Hb301 machines to measure hemoglobin levels in children in order to determine anemia prevalence using the WHO cut-offs: mild 10 ≤ hb < 11 g/dl; moderate 7 ≤ hb < 10 d/dl and severe hb < 7 g/dl. A finger prick will be used to obtain a drop of capillary blood that is placed on a cuvette and inserted in the Hemocue machine to obtain an on-the-spot assessment of hemoglobin levels. Population: A small number of children did not have hemoglobin measurements due to not wanting to have finger pricks or not being present for measurement.
  Participants
    number analyzed (Participants) | 200 | 278 | 478
    Child has no anemia | 61 | 86 | 147
    Child has anemia | 139 | 192 | 331
Number of children who consume a minimum acceptable diet [Count of Participants; unit: Participants] — A list-based recall will be used to assess dietary intake over the previous day. The 24-hour recall will be used to calculate minimum dietary diversity (MDD) (consuming 5 or more of 8 food groups and minimum meal frequency (MMF) (2x/day for breastfed infants 6-8 months; 3x/day for breastfed children 9-23 months; 4x/day for non-breastfed children 6-23 months). Children who meet the thresholds for both MDD and MMF are defined as consuming a MAD, based on the WHO/UNICEF IYCF indicator. Population: This measure was only for child participants
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Consumed minimum acceptable diet (MAD) | 29 | 25 | 54
    Did not consume minimum acceptable diet (MAD) | 176 | 258 | 434
Minimum dietary diversity consumed [Count of Participants; unit: Participants] — A 24-hour open dietary recall will be conducted with mothers to assess their child's dietary intake over the previous day. The 24-hour recall will be used to calculate the mean number of food groups (out of 8) consumed by the child over the previous day. Food groups include: breastmilk, grains, roots and tubers and plantains; pulses, nuts and seeds; dairy products; flesh foods; eggs; vitamin A rich fruits and vegetables; other fruit and vegetables. Population: We had missing data for one child
  Participants
    number analyzed (Participants) | 205 | 282 | 487
    Does not meet minimum dietary diversity | 159 | 224 | 383
    Meets minimum dietary diversity | 46 | 58 | 104
Minimum Meal Frequency [Count of Participants; unit: Participants] — Minimum meal frequency (MMF) is calculated based on the number of times the child is fed over the course of the day in night in the 24-hour dietary recall. Minimum meal frequency is met if the child is fed: 2x/day for breastfed infants 6-8.9 months; 3x/day for breastfed children 9-23.9 months; 4x/day for non-breastfed children 6-23.9 months. Population: This measure is for children participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Meets minimum meal frequency | 79 | 81 | 160
    Does not meet minimum meal frequency | 126 | 202 | 328
Bottle feeding 0-23 months [Count of Participants; unit: Participants] — Children 0-23 months of age who were fed from a bottle with a nipple during the previous day based on WHO IYCF indicators. Population: This measure is for children participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Child is bottle fed | 36 | 42 | 78
    Child is not bottle fed | 169 | 241 | 410
Egg and/or flesh food consumption [Count of Participants; unit: Participants] — Children 6-23 months of age who consumed egg and/or flesh food during the previous day. Population: This measure is for children participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Consumed eggs and/or flesh foods | 95 | 108 | 203
    Did not consume eggs and/or flesh foods | 110 | 175 | 285
Sweet beverage consumption [Count of Participants; unit: Participants] — Children 6-23 months of age who consumed a sweet beverage during the previous day. Population: This measure is for children participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Consumed sweet beverage | 93 | 134 | 227
    Did not consume sweet beverage | 112 | 149 | 261
Unhealthy food consumption [Count of Participants; unit: Participants] — Children 6-23 months of age who consumed selected sentinel unhealthy foods during the previous day. Unhealthy foods are defined based on the WHO IYCF indicator and includes: Selected sentinel unhealthy foods are:
  * Candies, chocolate and other sugar confections
  * Frozen treats like ice cream, gelato, sherbet, sorbet, popsicles or similar confections.
  * Cakes, pastries, sweet biscuits and other baked or fried confections
  * Chips, crisps, cheese puffs, French fries, fried dough, instant noodles and similar items Population: This measure is for children participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Consumed unhealthy food | 92 | 123 | 215
    Did not consume unhealthy food | 113 | 160 | 273
Zero vegetable or fruit consumption [Count of Participants; unit: Participants] — Children 6-23 months of age who did not consume any vegetables or fruits during the previous day. Population: This measure is for children participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Consumed vegetable and/or fruit | 49 | 88 | 137
    Did not consume vegetable and/or fruit | 156 | 195 | 351
Frequency of orange fruit and/or vegetable consumption in past 7 days [Mean (Standard Deviation); unit: number of times consumed] — The number of times the child has consumed orange fleshed fruits and/or vegetables over previous 7 days Population: This measure is for children participants only.
  number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 4.36 (4.24) | 3.96 (3.2) | 4.13 (3.7)
Animal-source food consumption over past 7 days [Mean (Standard Deviation); unit: Number of times consumed] — The number of times the child has consumed animal-source foods over the past 7 days Population: This measure is for children participants only.
  Number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 2.51 (2.86) | 2.75 (3.28) | 2.65 (3.11)
Leafy green consumption over past 7 days [Mean (Standard Deviation); unit: Number of times consumed] — The number of times the child has consumed leafy greens over the past 7 days Population: This measure is for children participants only.
  Number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 0.88 (1.93) | 0.77 (1.69) | 0.81 (1.79)
Thick porridge consumption [Mean (Standard Deviation); unit: Number of times consumed] — The number of times the child consumed thick porridge over the past 7 days Population: This measure is for children participants only.
  Number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 8.76 (9.84) | 10.93 (10.95) | 9.96 (10.5)
Consumption of porridge mixed with nutrient-rich food over past 7 days [Mean (Standard Deviation); unit: Number of times consumed] — The number of times the child was fed porridge mixed with other nutrient-rich foods over the past 7 days Population: This measure is for children participants only.
  Number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 3.62 (5.77) | 3.35 (5.14) | 3.46 (5.4)
Consumption of sugary foods over past 7 days [Mean (Standard Deviation); unit: Number of times consumed] — The number of times the child consumed sugary foods over the past 7 days Population: This measure is for children participants only.
  Number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 3.41 (3.34) | 3.41 (3.36) | 3.41 (3.35)
Consumption of fried foods over past 7 days [Mean (Standard Deviation); unit: Number of times consumed] — The number of times the child was fed fried foods over the past 7 days Population: This measure is for children participants only.
  Number of times consumed
    number analyzed (Participants) | 205 | 283 | 488
    (all) | 1.17 (2.42) | 0.94 (2.13) | 1.03 (2.26)
Mother's beliefs regarding infant and young child feeding practices [Count of Participants; unit: Participants] — Mother's beliefs about whether they should feed their young children leafy greens, animal-source foods, multiple times per day, orange fleshed fruits and vegetables (vitamin A rich), limiting sweets, providing clear or liquid porridge, handwashing, continuing to breastfeed after 6 months, and feeding the child a variety of foods at each meal. Scale is: strongly agree, agree, neutral, disagree and strongly disagree. Population: This measure is for mother participants only.
  Participants
    number analyzed (Participants) | 205 | 283 | 488
    Leafy greens will provide my baby with important nutrients: Strongly agree | 68 | 86 | 154
    Leafy greens will provide my baby with important nutrients: Agree | 86 | 111 | 197
    Leafy greens will provide my baby with important nutrients: Neutral (neither agree or disagree) | 28 | 61 | 89
    Leafy greens will provide my baby with important nutrients: Disagree | 22 | 17 | 39
    Leafy greens will provide my baby with important nutrients: Strongly disagree | 1 | 8 | 9
    Eating animal source foods can prevent anemia: Strongly agree | 88 | 124 | 212
    Eating animal source foods can prevent anemia: Agree | 95 | 121 | 216
    Eating animal source foods can prevent anemia: Neutral (neither agree or disagree) | 16 | 21 | 37
    Eating animal source foods can prevent anemia: Disagree | 6 | 15 | 21
    Eating animal source foods can prevent anemia: Strongly disagree | 0 | 2 | 2
    Feeding my baby multiple times a day is important for his/her growth and development: Strongly agree | 74 | 96 | 170
    Feeding my baby multiple times a day is important for his/her growth and development: Agree | 85 | 111 | 196
    Feeding my baby multiple times a day is important for his/her growth and development: Neutral (neither agree or disagree) | 8 | 16 | 24
    Feeding my baby multiple times a day is important for his/her growth and development: Disagree | 30 | 47 | 77
    Feeding my baby multiple times a day is important for his/her growth and development: Strongly disagree | 8 | 13 | 21
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Strongly agree | 97 | 141 | 238
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Agree | 97 | 131 | 228
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Neutral (neither agree or disagree) | 10 | 8 | 18
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Disagree | 1 | 3 | 4
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Strongly disagree | 0 | 0 | 0
    It is important to limit the amount of sweet and fried foods my baby consumes: Strongly agree | 80 | 98 | 178
    It is important to limit the amount of sweet and fried foods my baby consumes: Agree | 80 | 103 | 183
    It is important to limit the amount of sweet and fried foods my baby consumes: Neutral (neither agree or disagree) | 8 | 27 | 35
    It is important to limit the amount of sweet and fried foods my baby consumes: Disagree | 27 | 35 | 62
    It is important to limit the amount of sweet and fried foods my baby consumes: Strongly disagree | 10 | 20 | 30
    Clear or liquid porridge nourishes my baby: Strongly agree | 97 | 128 | 225
    Clear or liquid porridge nourishes my baby: Agree | 102 | 147 | 249
    Clear or liquid porridge nourishes my baby: Neutral (neither agree or disagree) | 3 | 3 | 6
    Clear or liquid porridge nourishes my baby: Disagree | 3 | 4 | 7
    Clear or liquid porridge nourishes my baby: Strongly disagree | 0 | 1 | 1
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Strongly agree | 127 | 180 | 307
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Agree | 69 | 90 | 159
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Neutral (neither agree or disagree) | 1 | 2 | 3
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Disagree | 5 | 6 | 11
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Strongly disagree | 3 | 5 | 8
    After six months, breast milk nourishes my baby: Strongly agree | 10 | 12 | 22
    After six months, breast milk nourishes my baby: Agree | 10 | 22 | 32
    After six months, breast milk nourishes my baby: Neutral (neither agree or disagree) | 0 | 2 | 2
    After six months, breast milk nourishes my baby: Disagree | 93 | 100 | 193
    After six months, breast milk nourishes my baby: Strongly disagree | 92 | 147 | 239
Father's beliefs regarding infant and young child feeding practices [Count of Participants; unit: Participants] — Measure Description: Father's beliefs about whether they should feed their young children leafy greens, animal-source foods, multiple times per day, orange fleshed fruits and vegetables (vitamin A rich), limiting sweets, providing clear or liquid porridge, handwashing, continuing to breastfeed after 6 months, and feeding the child a variety of foods at each meal. Scale is: strongly agree, agree, neutral, disagree and strongly disagree Population: Few of the fathers included in the triad were available (because they were working in farming fields or working outside the household in other occupations) to complete the surveys asking about their infant and young child feeding knowledge, attitudes and beliefs. However, these fathers still received the intervention (if in the experimental group).
  Participants
    number analyzed (Participants) | 45 | 66 | 111
    Leafy greens will provide my baby with important nutrients: Strongly agree | 23 | 20 | 43
    Leafy greens will provide my baby with important nutrients: Agree | 21 | 36 | 57
    Leafy greens will provide my baby with important nutrients: Neutral (neither agree or disagree) | 1 | 9 | 10
    Leafy greens will provide my baby with important nutrients: Disagree | 0 | 0 | 0
    Leafy greens will provide my baby with important nutrients: Strongly disagree | 0 | 1 | 1
    Eating animal source foods can prevent anemia: Strongly agree | 22 | 16 | 38
    Eating animal source foods can prevent anemia: Agree | 22 | 41 | 63
    Eating animal source foods can prevent anemia: Neutral (neither agree or disagree) | 0 | 5 | 5
    Eating animal source foods can prevent anemia: Disagree | 1 | 3 | 4
    Eating animal source foods can prevent anemia: Strongly disagree | 0 | 1 | 1
    Feeding my baby multiple times a day is important for his/her growth and development: Strongly agree | 16 | 15 | 31
    Feeding my baby multiple times a day is important for his/her growth and development: Agree | 17 | 31 | 48
    Feeding my baby multiple times a day is important for his/her growth and development: Neutral (neither agree or disagree) | 3 | 8 | 11
    Feeding my baby multiple times a day is important for his/her growth and development: Disagree | 7 | 11 | 18
    Feeding my baby multiple times a day is important for his/her growth and development: Strongly disagree | 2 | 1 | 3
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Strongly agree | 25 | 21 | 46
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Agree | 18 | 42 | 60
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Neutral (neither agree or disagree) | 2 | 3 | 5
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Disagree | 0 | 0 | 0
    Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Strongly disagree | 0 | 0 | 0
    It is important to limit the amount of sweet and fried foods my baby consumes: Strongly agree | 21 | 15 | 36
    It is important to limit the amount of sweet and fried foods my baby consumes: Agree | 17 | 33 | 50
    It is important to limit the amount of sweet and fried foods my baby consumes: Neutral (neither agree or disagree) | 2 | 5 | 7
    It is important to limit the amount of sweet and fried foods my baby consumes: Disagree | 3 | 8 | 11
    It is important to limit the amount of sweet and fried foods my baby consumes: Strongly disagree | 2 | 5 | 7
    Clear or liquid porridge nourishes my baby: Strongly agree | 22 | 21 | 43
    Clear or liquid porridge nourishes my baby: Agree | 23 | 42 | 65
    Clear or liquid porridge nourishes my baby: Neutral (neither agree or disagree) | 0 | 3 | 3
    Clear or liquid porridge nourishes my baby: Disagree | 0 | 0 | 0
    Clear or liquid porridge nourishes my baby: Strongly disagree | 0 | 0 | 0
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Strongly agree | 28 | 33 | 61
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Agree | 17 | 31 | 48
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Neutral (neither agree or disagree) | 0 | 1 | 1
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Disagree | 0 | 1 | 1
    Washing hands with soap before & after cooking, eating, etc. can help prevent illness: Strongly disagree | 0 | 0 | 0
    After six months, breast milk nourishes my baby: Strongly agree | 8 | 5 | 13
    After six months, breast milk nourishes my baby: Agree | 5 | 10 | 15
    After six months, breast milk nourishes my baby: Neutral (neither agree or disagree) | 3 | 4 | 7
    After six months, breast milk nourishes my baby: Disagree | 13 | 31 | 44
    After six months, breast milk nourishes my baby: Strongly disagree | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Who Consume a Minimum Acceptable Diet
Description: The minimum acceptable diet indicator will be used to assess diet quality in children. A list-based recall will be used to assess dietary intake over the previous day. The 24-hour recall will be used to calculate minimum dietary diversity (MDD) (consuming 5 or more of 8 food groups (breast milk; grains, roots, tubers and plantains; pulses (beans, peas, lentils), nuts and seeds; dairy products (milk, infant formula, yogurt, cheese); flesh foods (meat, fish, poultry, organ meats); eggs; vitamin A rich fruits and vegetables; other fruit and vegetables) and minimum meal frequency (MMF) (2x/day for breastfed infants 6-8 months; 3x/day for breastfed children 9-23 months; 4x/day for non-breastfed children 6-23 months). Children who meet the thresholds for both MDD and MMF are defined as consuming a MAD, based on the WHO/UNICEF IYCF indicator.
Time Frame: At study completion, an average of 4 months after baseline
Population: Children in both the control group and the intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 205 | 283
Participants
  Consumed minimum acceptable diet (MAD) | 67 | 92
  Did not consume minimum acceptable diet | 138 | 191
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority; p = 0.145, Regression, Logistic — The a priori threshold for statistical significance is <0.05. The p-value is for the intervention by time interaction; Odds Ratio (OR) = 0.9585, 95% CI 2-sided [0.4276 to 2.1485] — Odds of consuming a minimum acceptable diet in control group at endline
Statistical Analysis 2: Comparison: Infant and Young Child Feeding (IYCF) Voice Messaging Intervention; Test type: Superiority; p = 0.145, Regression, Logistic — The a priori threshold for statistical significance is <0.05. The p-value is for the intervention by time interaction; Odds Ratio (OR) = 0.9669, 95% CI 2-sided [0.43 to 2.1742] — Odds of consuming a minimum acceptable diet in intervention group at endline

2. Primary Outcome: Anemia Prevalence of Children
Description: Hemocue Hb301 machines to measure hemoglobin levels in children in order to determine anemia prevalence using the WHO cut-offs: mild 10 ≤ hb < 11 g/dl; moderate 7 ≤ hb < 10 d/dl and severe hb < 7 g/dl. A finger prick will be used to obtain a drop of capillary blood that is placed on a cuvette and inserted in the Hemocue machine to obtain an on-the-spot assessment of hemoglobin levels.
Time Frame: At study completion, an average of 4 months after baseline
Population: Children in both control and intervention group post intervention implementation. The number of children included in the sample is smaller than the participant flow module given that not all children completed the hemoglobin measurement due to not consenting to it or because the child was not present at the time of data collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 170 | 236
Participants
  Anemia | 123 | 154
  No anemia | 47 | 82
Statistical Analysis 1: Comparison: Control Group; Test type: Superiority; p = 0.179, Regression, Logistic — The a priori threshold for statistical significance is <0.05. The p-value is for the intervention by time interaction; Odds Ratio (OR) = 0.3084, 95% CI 2-sided [0.1977 to 0.481]
Statistical Analysis 2: Comparison: Infant and Young Child Feeding (IYCF) Voice Messaging Intervention; Test type: Superiority; p = 0.179, Regression, Logistic — The a priori threshold for statistical significance is <0.05. The p-value is for the intervention by time interaction; Odds Ratio (OR) = 0.438, 95% CI 2-sided [0.2983 to 0.6431]

3. Primary Outcome: Change in Percentage of Children Consuming a Minimum Acceptable Diet Between Baseline and Endline
Description: The change in percentage of children meeting the minimum acceptable diet indicator between baseline and endline will be used to assess diet quality in children. A list-based recall will be used to assess dietary intake over the previous day. The 24-hour recall will be used to calculate minimum dietary diversity (MDD) (consuming 5 or more of 8 food groups (breast milk; grains, roots, tubers and plantains; pulses (beans, peas, lentils), nuts and seeds; dairy products (milk, infant formula, yogurt, cheese); flesh foods (meat, fish, poultry, organ meats); eggs; vitamin A rich fruits and vegetables; other fruit and vegetables) and minimum meal frequency (MMF) (2x/day for breastfed infants 6-8 months; 3x/day for breastfed children 9-23 months; 4x/day for non-breastfed children 6-23 months). Children who meet the thresholds for both MDD and MMF are defined as consuming a MAD, based on the WHO/UNICEF IYCF indicator.
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Population: Analysis of children in control and intervention group, post-intervention implementation.
Measure: Number; unit: percent of participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 205 | 283
percent of participants | 18.5 | 23.7

4. Primary Outcome: Change in Percentage of Children With Anemia Between Baseline and Endline
Description: We will use Hemocue Hb301 machines to measure hemoglobin levels in children in order to determine anemia prevalence using the WHO cut-offs: mild 10 ≤ hb < 11 g/dl; moderate 7 ≤ hb < 10 d/dl and severe hb < 7 g/dl. A finger prick will be used to obtain a drop of capillary blood that is placed on a cuvette and inserted in the Hemocue machine to obtain an on-the-spot assessment of hemoglobin levels. The change in child anemia prevalence between baseline and endline will be examined (calculated as endline-baseline/baseline*100).
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Population: Children in control and intervention group, post-intervention implementation
Measure: Number; unit: percent of participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 170 | 236
percent of participants | 2.9 | -3.8

5. Secondary Outcome: Frequency of Child Consuming Key Foods in the Past 7 Days
Description: The frequency of the child consuming specific foods targeted in the intervention over the course of the previous week (7 days) will be assessed. More specifically, the number of times that the following foods have been consumed will be assessed: animal source foods, leafy greens, orange colored fruits and vegetables, thick porridge, porridge mixed with nutrient-rich foods, sweets and sugary drinks, fried foods.
Time Frame: At study completion, an average of 4 months after baseline
Population: We have some missing data for children at endline.
Measure: Mean (Standard Deviation); unit: Times key foods consumed in past 7 days
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 177 | 239
Times key foods consumed in past 7 days
  Frequency of consuming orange fruits and/or vegetables over past 7 days | 4.7 (2.85) | 4.97 (2.77)
  Frequency of consuming animal source foods over past 7 days | 4.40 (2.94) | 4.55 (2.93)
  Frequency of consuming leafy greens over past 7 days | 2.03 (2.79) | 2.05 (2.6)
  Frequency of consuming thick porridge over past 7 days | 8.88 (13.95) | 9.51 (14.31)
  Frequency of consuming porridge mixed with nutrient rich foods over past 7 days | 3.47 (4.49) | 3.51 (4.40)
  Frequency of consuming sugary foods over the past 7 days | 6.72 (5.25) | 6.52 (5.16)
  Frequency of consuming fried foods over the past 7 days | 1.77 (2.48) | 1.69 (2.52)

6. Secondary Outcome: Infant and Young Child Feeding (IYCF) Practices Indicators
Description: The WHO/UNICEF IYCF indicators will be used to assess feeding practices. Mothers will be asked about feeding practices as part of the household surveys. The indicators include: ever breastfed, early initiation of breastfeeding, exclusively breastfed for the first two days after birth, bottle feeding 0-23 months, continued breastfeeding 12-23 months, introduction of solid, semi-solid or soft foods 6-8 months, egg and/or flesh food consumption, sweet beverage consumption, unhealthy food consumption, and zero vegetable or fruit. The proportion of children being fed according to the detailed descriptions of these indicators will be assessed based on the WHO/UNICEF IYCF indicator manual.
Time Frame: At study completion, an average of 4 months after baseline
Population: We have missing data for some children at endline leading to a smaller sample size
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 205 | 283
Participants
  Bottle feeding: number analyzed (Participants) | 177 | 239
  Bottle feeding: Yes | 10 | 18
  Bottle feeding: No | 167 | 221
  Egg and/or flesh food consumption: Yes | 123 | 168
  Egg and/or flesh food consumption: No | 82 | 115
  Sweet beverage consumption: Yes | 93 | 178
  Sweet beverage consumption: No | 112 | 105
  Unhealthy food consumption: Yes | 107 | 156
  Unhealthy food consumption: No | 98 | 127
  Zero vegetable or fruit consumption: Yes | 25 | 25
  Zero vegetable or fruit consumption: No | 180 | 258

7. Secondary Outcome: Mothers and Fathers Infant and Young Child Feeding (IYCF) Knowledge, Attitudes, Norms and Intentions
Description: IYCF knowledge, attitudes, norms and intentions will be assessed using survey questions based on the components of the intervention. Both mothers and fathers will be asked the survey questions as part of the household survey. The questions are grounded in the theory of planned behavior and based on previously published IYCF knowledge, attitudes, norms and intentions questions. The questions have been pilot tested by the project PI.
Time Frame: At study completion, an average of 4 months after baseline
Population: We report the mothers' and fathers' beliefs related to infant and young child feeding practices. There is some missing data which is why we have a smaller sample size. For fathers, very few were present to participate in survey questions. However, fathers in experimental group still received the intervention if they did not participate in the survey.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Mothers in Triad; Control Group: Fathers in Triad: The control group will not receive any intervention. After the endline data collection is completed, the intervention will be delivered to the control group.
- Infant and Young Child Feeding (IYCF) Voice Messaging Intervention: Mothers in Triad; Infant and Young Child Feeding (IYCF) Voice Messaging Intervention: Fathers in Triad: The voice messaging intervention group will receive voice/text messages for a period of 16 weeks.
  Infant and young child feeding voice messaging intervention: A mobile voice and text messaging intervention aimed at improving IYCF practices will be delivered to mothers and fathers with young children (6-23 months). A total of 16 voice and text message, with the same content, will be sent over a 16-week period (1 voice + 1 text messages (with same content) per week x 16 weeks). Two types of messages will be included: 1) eight scripted and 2) eight unscripted messages from positive deviants. The content of the messages include: breastfeeding until two years of age, consuming a variety of foods within a given meal, the consistency of porridge (thick rather than thin), limiting sweets and fried foods, the importance of animal source foods, consuming vitamin A rich fruits and vegetables, consuming leafy greens, handwashing and feeding infants and young children fruits and vegetables produced by the household.
Arm/Group | Control Group: Mothers in Triad | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention: Mothers in Triad | Control Group: Fathers in Triad | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention: Fathers in Triad
Number analyzed (Participants) | 177 | 239 | 28 | 48
Participants
  Leafy greens will provide my baby with important nutrients: Strongly agree | 93 | 113 | 15 | 25
  Leafy greens will provide my baby with important nutrients: Agree | 69 | 101 | 12 | 22
  Leafy greens will provide my baby with important nutrients: Neutral (neither agree or disagree) | 11 | 16 | 1 | 1
  Leafy greens will provide my baby with important nutrients: Disagree | 4 | 5 | 0 | 0
  Leafy greens will provide my baby with important nutrients: Strongly disagree | 0 | 4 | 0 | 0
  Eating animal source foods can prevent anemia: Strongly agree | 86 | 121 | 15 | 23
  Eating animal source foods can prevent anemia: Agree | 83 | 111 | 13 | 24
  Eating animal source foods can prevent anemia: Neutral (neither agree or disagree) | 6 | 2 | 0 | 1
  Eating animal source foods can prevent anemia: Disagree | 1 | 4 | 0 | 0
  Eating animal source foods can prevent anemia: Strongly disagree | 1 | 1 | 0 | 0
  Feeding my baby multiple times a day is important for his/her growth and development: Strongly agree | 76 | 103 | 15 | 23
  Feeding my baby multiple times a day is important for his/her growth and development: Agree | 74 | 83 | 9 | 20
  Feeding my baby multiple times a day is important for his/her growth and development: Neutral (neither agree or disagree) | 6 | 13 | 1 | 0
  Feeding my baby multiple times a day is important for his/her growth and development: Disagree | 16 | 36 | 3 | 5
  Feeding my baby multiple times a day is important for his/her growth and development: Strongly disagree | 5 | 4 | 0 | 0
  Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Strongly agree | 86 | 126 | 16 | 26
  Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Agree | 89 | 110 | 11 | 21
  Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Neutral (neither agree or disagree) | 2 | 3 | 1 | 1
  Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Disagree | 0 | 0 | 0 | 0
  Feeding my baby orange fruits and vegetables can help their eye health and prevent illness: Strongly disagree | 0 | 0 | 0 | 0
  It is important to limit the amount of sweet and fried foods my baby consumes: Strongly agree | 55 | 58 | 13 | 21
  It is important to limit the amount of sweet and fried foods my baby consumes: Agree | 67 | 89 | 7 | 14
  It is important to limit the amount of sweet and fried foods my baby consumes: Neutral (neither agree or disagree) | 20 | 24 | 2 | 2
  It is important to limit the amount of sweet and fried foods my baby consumes: Disagree | 17 | 38 | 3 | 6
  It is important to limit the amount of sweet and fried foods my baby consumes: Strongly disagree | 18 | 30 | 3 | 5
  Clear or liquid porridge nourishes my baby: Strongly agree | 63 | 93 | 9 | 24
  Clear or liquid porridge nourishes my baby: Agree | 89 | 120 | 18 | 22
  Clear or liquid porridge nourishes my baby: Neutral (neither agree or disagree) | 12 | 4 | 0 | 1
  Clear or liquid porridge nourishes my baby: Disagree | 8 | 17 | 1 | 1
  Clear or liquid porridge nourishes my baby: Strongly disagree | 5 | 5 | 0 | 0
  Washing my hands with soap before and after cooking, eating, etc. can help prevent illness: Strongly agree | 104 | 144 | 16 | 29
  Washing my hands with soap before and after cooking, eating, etc. can help prevent illness: Agree | 73 | 92 | 12 | 19
  Washing my hands with soap before and after cooking, eating, etc. can help prevent illness: Neutral (neither agree or disagree) | 0 | 0 | 0 | 0
  Washing my hands with soap before and after cooking, eating, etc. can help prevent illness: Disagree | 0 | 1 | 0 | 0
  Washing my hands with soap before and after cooking, eating, etc. can help prevent illness: Strongly disagree | 0 | 2 | 0 | 0
  After six months, breast milk nourishes my baby: Strongly agree | 23 | 21 | 6 | 10
  After six months, breast milk nourishes my baby: Agree | 36 | 36 | 6 | 13
  After six months, breast milk nourishes my baby: Neutral (neither agree or disagree) | 1 | 2 | 9 | 12
  After six months, breast milk nourishes my baby: Disagree | 49 | 75 | 7 | 13
  After six months, breast milk nourishes my baby: Strongly disagree | 68 | 105 | 0 | 0

8. Secondary Outcome: Number of Children Consuming Minimum Meal Frequency
Description: Minimum meal frequency of (semi) solid or soft foods is assessed by examining the proportion of young children consuming foods: 2x/day for breastfed infants 6-8 months; 3x/day for breastfed children 9-23 months; 4x/day for non-breastfed children 6-23 months)
Time Frame: At study completion, an average of 4 months after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 205 | 283
Participants
  Consumed minimum meal frequency | 121 | 142
  Did not consume minimum meal frequency | 84 | 141
Statistical Analysis 1: Comparison: Control Group vs Infant and Young Child Feeding (IYCF) Voice Messaging Intervention; Test type: Superiority; p = 0.054, Chi-squared — A priori threshold for statistical significance <0.05

9. Secondary Outcome: Number of Children Consuming Minimum Dietary Diversity
Description: The proportion of young children consuming 5 or more of 8 food groups (breast milk; grains, roots, tubers and plantains; pulses (beans, peas, lentils), nuts and seeds; dairy products (milk, infant formula, yogurt, cheese); flesh foods (meat, fish, poultry, organ meats); eggs; vitamin A rich fruits and vegetables; other fruit and vegetables)
Time Frame: At study completion, an average of 4 months after baseline
Population: Population includes children in the study. We had missing data for some children at endline, which is the reason for the smaller sample size
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 176 | 238
Participants
  Did not meet minimum dietary diversity | 85 | 102
  Met minimum dietary diversity | 91 | 136
Statistical Analysis 1: Comparison: Control Group vs Infant and Young Child Feeding (IYCF) Voice Messaging Intervention; Test type: Superiority; p = 0.65, Chi-squared — A priori threshold for statistical significance <0.05

10. Secondary Outcome: Percent Change in Frequency of Consuming Key Foods in the Past 7 Days
Description: The percent change (calculated as endline-baseline/baseline) in the frequency of consuming specific foods targeted in the intervention over the course of the previous week (7 days) will be assessed between baseline and endline. More specifically, the number of times that the following foods have been consumed will be assessed: animal source foods, leafy greens, orange colored fruits and vegetables, thick porridge, porridge mixed with nutrient-rich foods, sweets and sugary drinks, fried foods.
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Population: We have missing data for some variables, which is why there are smaller numbers. In addition, we had participants who consumed 0 servings at baseline which led to this variable not being able to be calculated for them.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 177 | 239
percent change
  Percent change in frequency of consuming orange fruits and/or vegetables over past 7 days: number analyzed (Participants) | 141 | 194
  Percent change in frequency of consuming orange fruits and/or vegetables over past 7 days | 44.4 (161.4) | 51.6 (157.3)
  Percent change in frequency of consuming animal source foods over past 7 days: number analyzed (Participants) | 101 | 137
  Percent change in frequency of consuming animal source foods over past 7 days | 71.6 (176.5) | 46.1 (150.7)
  Percent change in frequency of consuming leafy greens over past 7 days: number analyzed (Participants) | 49 | 63
  Percent change in frequency of consuming leafy greens over past 7 days | 31.1 (170.8) | 56.7 (208.5)
  Percent change in frequency of consuming thick porridge over past 7 days: number analyzed (Participants) | 45 | 46
  Percent change in frequency of consuming thick porridge over past 7 days | 5.2 (268.5) | 15.0 (288.3)
  Percent change in frequency of consuming porridge mixed with nutrient rich foods over past 7 days: number analyzed (Participants) | 109 | 154
  Percent change in frequency of consuming porridge mixed with nutrient rich foods over past 7 days | 52.0 (282.8) | 48.6 (270.9)
  Percent change in frequency of consuming sugary foods over the past 7 days: number analyzed (Participants) | 101 | 151
  Percent change in frequency of consuming sugary foods over the past 7 days | 90.7 (276.8) | 117.2 (315.0)
  Percent change in frequency of consuming fried foods over the past 7 days: number analyzed (Participants) | 52 | 67
  Percent change in frequency of consuming fried foods over the past 7 days | 17.7 (187.4) | -35.1 (123.8)

11. Secondary Outcome: Change in Percentage of Children Meeting Recommended Infant and Young Child Feeding (IYCF) Practices Indicators
Description: The change in percentage of children being fed according to the recommended IYCF practices between baseline and endline. The WHO/UNICEF IYCF indicators will be used to assess feeding practices. Mothers will be asked about feeding practices as part of the household surveys. The indicators include: ever breastfed, early initiation of breastfeeding, exclusively breastfed for the first two days after birth, bottle feeding 0-23 months, continued breastfeeding 12-23 months, introduction of solid, semi-solid or soft foods 6-8 months, egg and/or flesh food consumption, sweet beverage consumption, unhealthy food consumption, and zero vegetable or fruit.
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Population: We have some missing data. In these cases, the sample size is lower than the total sample.
Measure: Number; unit: percent of participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 205 | 283
percent of participants
  Change in percentage of children bottle fed: number analyzed (Participants) | 177 | 239
  Change in percentage of children bottle fed | -11.9 | -7.3
  Change in percentage of children fed egg and/or flesh food consumption | 13.7 | 21.2
  Change in percentage of children fed sweet beverage consumption | 17.1 | 15.6
  Change in percentage of children fed unhealthy food | 7.3 | 11.7
  Change in percentage of children fed zero vegetable or fruit | -11.7 | -22.3

12. Secondary Outcome: Change in Percentage of Children Meeting Minimum Meal Frequency Indicator
Description: The change in the percentage of children meeting the minimum meal frequency (MMF) indicator between baseline and endline will be assessed. Minimum meal frequency of (semi) solid or soft foods is assessed by examining the proportion of young children consuming foods: 2x/day for breastfed infants 6-8 months; 3x/day for breastfed children 9-23 months; 4x/day for non-breastfed children 6-23 months.
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Measure: Number; unit: percent of participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 205 | 283
percent of participants | 20.5 | 21.6

13. Secondary Outcome: Change in Percentage of Children Meeting Minimum Dietary Diversity
Description: The change in the percentage of young children consuming 5 or more of 8 food groups (breast milk; grains, roots, tubers and plantains; pulses (beans, peas, lentils), nuts and seeds; dairy products (milk, infant formula, yogurt, cheese); flesh foods (meat, fish, poultry, organ meats); eggs; vitamin A rich fruits and vegetables; other fruit and vegetables) between baseline and endline.
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Population: We have some missing data for some children. Numbers reported are for endline time point.
Measure: Number; unit: percent of participants
Arm/Group | Control Group | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention
Number analyzed (Participants) | 176 | 238
percent of participants | 29.3 | 36.6

14. Secondary Outcome: Change in Percentage of Mothers and Fathers Infant and Young Child Feeding (IYCF) Knowledge, Attitudes, Norms and Intentions
Description: The change in percentage of mothers/fathers with specific IYCF knowledge, attitudes, norms and intentions between baseline and endline will be assessed using survey questions based on the components of the intervention. Mothers will be asked the survey questions as part of the household survey. The questions are grounded in the theory of planned behavior and based on previously published IYCF knowledge, attitudes, norms and intentions questions.
Time Frame: Between baseline and study completion, an average of 4 months after baseline
Population: Mother's of children included in study sample. We have some missing data related to mother's IYCF beliefs. For this reason, the sample size is smaller than the whole sample.
Measure: Number; unit: percent of participants
Groups:
- Infant and Young Child Feeding (IYCF) Voice Messaging: Fathers in Triad: The voice messaging intervention group will receive voice/text messages for a period of 16 weeks.
  Infant and young child feeding voice messaging intervention: A mobile voice and text messaging intervention aimed at improving IYCF practices will be delivered to mothers and fathers with young children (6-23 months). A total of 16 voice and text message, with the same content, will be sent over a 16-week period (1 voice + 1 text messages (with same content) per week x 16 weeks). Two types of messages will be included: 1) eight scripted and 2) eight unscripted messages from positive deviants. The content of the messages include: breastfeeding until two years of age, consuming a variety of foods within a given meal, the consistency of porridge (thick rather than thin), limiting sweets and fried foods, the importance of animal source foods, consuming vitamin A rich fruits and vegetables, consuming leafy greens, handwashing and feeding infants and young children fruits and vegetables produced by the household.
Arm/Group | Control Group: Mothers in Triad | Infant and Young Child Feeding (IYCF) Voice Messaging Intervention: Mothers in Triad | Control Group: Fathers in Triad | Infant and Young Child Feeding (IYCF) Voice Messaging: Fathers in Triad
Number analyzed (Participants) | 177 | 239 | 28 | 48
percent of participants
  Change in percentage of mothers/fathers strongly agreeing leafy greens provide important nutrients | 19.4 | 16.9 | 2.5 | 21.8
  Change in percentage of mothers/fathers strongly agreeing animal source foods can prevent anemia | 5.7 | 6.8 | 4.7 | 23.7
  Change in percentage of mothers/fathers strongly agree feeding baby multiple times/day is important | 6.8 | 9.2 | 18.0 | 25.2
  Change in percentage of mothers/fathers strongly agree feeding orange fruits/vegetables is important | 1.3 | 2.9 | 1.6 | 22.4
  Change in percentage of mothers/fathers strongly agree that limiting amount of sweet and fried foods | -8.0 | -10.4 | -0.2 | 21.0
  Change in percentage of mothers/fathers that strongly agree clear or liquid porridge nourishes baby | -11.7 | -6.3 | -16.8 | 18.2
  Change in percentage of mothers/fathers that strongly agree about importance of washing hands | -3.2 | -3.4 | -5.1 | 10.4
  Change in percentage of mothers/fathers that believe breast milk nourishes baby after 6 mths | 8.1 | 4.6 | 3.7 | 13.3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the intervention (approximately 6 months (inclusive of baseline and endline data collection)) for the triad (mothers, fathers, children).
Description: The definition of adverse event does not differ from the definition provided by clinicaltrials.gov
Groups:
- Control Group - Children: The control group will not receive any intervention. After the endline data collection is completed, the intervention will be delivered to the control group. This group includes the children participants.
- Control Group - Mothers: The control group will not receive any intervention. After the endline data collection is completed, the intervention will be delivered to the control group. This group includes the mother participants.
- Control Group - Fathers: The control group will not receive any intervention. After the endline data collection is completed, the intervention will be delivered to the control group. This group includes the father participants.
- Infant and Young Child Feeding - (IYCF) Voice Messaging Intervention - Children: The voice messaging intervention group will receive voice/text messages for a period of 16 weeks.
  Infant and young child feeding voice messaging intervention: A mobile voice and text messaging intervention aimed at improving IYCF practices will be delivered to mothers and fathers with young children (6-23 months). A total of 16 voice and text message, with the same content, will be sent over a 16-week period (1 voice + 1 text messages (with same content) per week x 16 weeks). Two types of messages will be included: 1) eight scripted and 2) eight unscripted messages from positive deviants. The content of the messages include: breastfeeding until two years of age, consuming a variety of foods within a given meal, the consistency of porridge (thick rather than thin), limiting sweets and fried foods, the importance of animal source foods, consuming vitamin A rich fruits and vegetables, consuming leafy greens, handwashing and feeding infants and young children fruits and vegetables produced by the household. This group includes the children participants.
- Infant and Young Child Feeding - (IYCF) Voice Messaging Intervention - Mothers: The voice messaging intervention group will receive voice/text messages for a period of 16 weeks.
  Infant and young child feeding voice messaging intervention: A mobile voice and text messaging intervention aimed at improving IYCF practices will be delivered to mothers and fathers with young children (6-23 months). A total of 16 voice and text message, with the same content, will be sent over a 16-week period (1 voice + 1 text messages (with same content) per week x 16 weeks). Two types of messages will be included: 1) eight scripted and 2) eight unscripted messages from positive deviants. The content of the messages include: breastfeeding until two years of age, consuming a variety of foods within a given meal, the consistency of porridge (thick rather than thin), limiting sweets and fried foods, the importance of animal source foods, consuming vitamin A rich fruits and vegetables, consuming leafy greens, handwashing and feeding infants and young children fruits and vegetables produced by the household. This group includes the mother participants.
- Infant and Young Child Feeding - (IYCF) Voice Messaging Intervention - Fathers: The voice messaging intervention group will receive voice/text messages for a period of 16 weeks.
  Infant and young child feeding voice messaging intervention: A mobile voice and text messaging intervention aimed at improving IYCF practices will be delivered to mothers and fathers with young children (6-23 months). A total of 16 voice and text message, with the same content, will be sent over a 16-week period (1 voice + 1 text messages (with same content) per week x 16 weeks). Two types of messages will be included: 1) eight scripted and 2) eight unscripted messages from positive deviants. The content of the messages include: breastfeeding until two years of age, consuming a variety of foods within a given meal, the consistency of porridge (thick rather than thin), limiting sweets and fried foods, the importance of animal source foods, consuming vitamin A rich fruits and vegetables, consuming leafy greens, handwashing and feeding infants and young children fruits and vegetables produced by the household. This group includes the father participants.
Arm/Group | Control Group - Children | Control Group - Mothers | Control Group - Fathers | Infant and Young Child Feeding - (IYCF) Voice Messaging Intervention - Children | Infant and Young Child Feeding - (IYCF) Voice Messaging Intervention - Mothers | Infant and Young Child Feeding - (IYCF) Voice Messaging Intervention - Fathers
All-Cause Mortality (participants affected / at risk) | 0/205 | 0/205 | 0/45 | 0/283 | 0/283 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/205 | 0/205 | 0/45 | 0/283 | 0/283 | 0/66
Other Adverse Events (participants affected / at risk) | 0/205 | 0/205 | 0/45 | 0/283 | 0/283 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT05374837/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT05374837/SAP_001.pdf
  • Informed Consent Form (2022-07-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT05374837/ICF_002.pdf